CLINICAL TRIAL: NCT01138930
Title: Effect of Berberine on Hormonal and Metabolic Features in Obese Women With PCOS
Brief Title: Effect of Berberine on Hormonal and Metabolic Features in Obese Women With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Chairman Dept Obs & Gyn, First Affiliated Hospital, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: berberine2010
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Polycystic Ovary Syndrome; Obesity
Keywords: Polycystic Ovary Syndrome; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Berberine (Experimental)
  Interventions: Drug: Berberine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine — 1.5g daily for 3 month
  Arms: Berberine
Drug: Placebo — placebo daily
  Arms: Placebo

SUMMARY:
Berberine has showed effective in lowering blood sugar levels in db/db mice and anti-dyslipidemia in human.Studies on the effect of berberine on metabolic and hormonal features of women with polycystic ovary syndrome (PCOS) are lacking.The objective of this study is to examine the effect of Berberine metabolic and hormonal parameters and insulin resistance in obese patients with PCOS.

ELIGIBILITY:
Inclusion Criteria

1. Age of women between 18 and 35 years.
2. Confirmed diagnosis of PCOS according to the modified Rotterdam criteria and all subjects must have anovulation plus either polycystic ovaries and/or hyperandrogenism.
3. Body mass index (BMI) equal to or greater than 23 kg/m2.
4. With no desire of children within 6 month. PCOS is defined by the modified Rotterdam criteria: oligomenorrhea or amenorrhea, together with presence of ≥12 antral follicles (≤9mm) and/or ovarian volume >10 ml on transvaginal scanning, and/or clinical/biochemical hyperandrogenism. Oligomenorrhea is defined as an intermenstrual interval >35 days and <8 menstrual bleedings in the past year. Amenorrhea is defined as an intermenstrual interval >90 days. Clinical hyperandrogenism in China Mainland is defined as a Ferriman-Gallwey (FG) score ≥5.

Exclusion criteria are

1. Use of hormonal drugs or other medications including Chinese Herbal prescriptions in the past 3 months.
2. Patients with other endocrine disorders including 21-hydroxylase deficiency, hyperprolactinemia, uncorrected thyroid disease, suspected Cushing's syndrome
3. Patients with known sever organ dysfunction or mental illness.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Whole body insulin action | 3 months
  Glucose Disposal Rate measured by hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
Oral glucose tolerance test (OGTT) | 3 months
Ovarian androgen biosynthesis | 3 months
Hormonal profile | 3 months
Fasting lipid metabolic profile | 3 months
Renal and liver function tests | 3 months
Adverse events | 3 months
6) Weight, waist/hip circumference, blood pressure, F-G score and acne before and after treatment. | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Lihui Hou, MD., Study Chair — The First Affliated Hospital,Heilongjiang University of Chinese Medicine .; Xiaoke Wu, MD.PhD., Study Chair — The First Affliated Hospital,Heilongjiang University of Chinese Medicine
Locations (4):
- China (4):
  - Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Forth Affiliated Hospital of Harbin Medcal University, Harbin, Heilongjiang
  - Department of Obstetrics and Gynecology,First Affliated Hospital,Heilongjiang University of Chinese Medicine ., Harbin, Heilongjiang

REFERENCES:
- [Derived] Zhang Y, Sun J, Zhang YJ, Chai QY, Zhang K, Ma HL, Wu XK, Liu JP. The effect of berberine on insulin resistance in women with polycystic ovary syndrome: detailed statistical analysis plan (SAP) for a multicenter randomized controlled trial. Trials. 2016 Oct 21;17(1):512. doi: 10.1186/s13063-016-1633-5. PMID 27769284
- [Derived] Li Y, Ma H, Zhang Y, Kuang H, Ng EH, Hou L, Wu X. Effect of berberine on insulin resistance in women with polycystic ovary syndrome: study protocol for a randomized multicenter controlled trial. Trials. 2013 Jul 18;14:226. doi: 10.1186/1745-6215-14-226. PMID 23866924